CLINICAL TRIAL: NCT01486563
Title: Effect of Hydroxyethyl Starch on Renal Handling of Sodium and Water, Vasoactive Hormones,Biomarkers and the Circulatory System in Patients Undergoing Radical Prostatectomy
Brief Title: Hydroxyethyl Starch and Renal Function After Radical Prostatectomy
Acronym: VORA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Principal Investigator, Erling Bjerregaard Pedersen, Professor, Regional Hospital Holstebro
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: ASK-2-2011
Record Dates: First submitted 2011-12-04; First posted 2011-12-06 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — HES 130-0.4; Hydroxyethyl Starch Derivatives; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Voluven (Hydroxyethyl starch 130/0,4) (Active Comparator): Patients undergoing radical prostatectomy will receive either fluid therapy with active comparator (Voluven) or placebo (Sodium Chloride)
  Interventions: Drug: Voluven (Hydroxyethyl starch 130/0,4)
- Sodium Chloride 9 mg/ml (Placebo Comparator): Patients undergoing radical prostatectomy will receive either fluid therapy with active comparator (Voluven) or placebo (Sodium Chloride)
  Interventions: Drug: Sodium Chloride 9 mg/ml

INTERVENTIONS:
Drug: Voluven (Hydroxyethyl starch 130/0,4) — 7,5 ml/kg in the first hour and then 5 ml/kg
  Other Names: Voluven; Venofundin; Hydroxyethyl starch
  Arms: Voluven (Hydroxyethyl starch 130/0,4)
Drug: Sodium Chloride 9 mg/ml — 7,5 ml/kg in the first hour and then 5 ml/kg
  Other Names: Istone saline solution
  Arms: Sodium Chloride 9 mg/ml

SUMMARY:
The purpose of this project is to investigate if hydroxyethyl starch (HES) is potential nephrotoxic and examine the effects on the circulation and kidneys during administration of HES during surgery.

DETAILED DESCRIPTION:
Hydroxyethyl starch (HES) is widely used in hospitals to maintain circulation in critically ill patients. In recent years studies have raised suspicion that HES is nephrotoxic. So far acute kidney injury has been diagnosed based on creatinine measurements, but new technology allows for earlier diagnosis using measurements of biomarkers in urine.

The purpose of this project is to investigate HES's potential toxicity and effects on the circulation and kidneys using measurements of biomarkers specific for toxicity and for the sodium/water balance in the urine and by measurements of vasoactive hormones in the blood after administration of HES 130/0.4

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Males
* Indication for radical prostatectomy

Exclusion Criteria:

* Blood donation within the last month
* Lack of wish to participate
* eGFR< 15ml/min

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
u-NGAL | 2-4 hours
  The main objective for the trial (only patients undergoing elective radical prostatectomy) is to measure the effect of hydroxyethyl starch on u-NGAL, which is a biomarker of nephrotoxicity

SECONDARY OUTCOMES:
u-Kim 1, u- FABP | 2-4 hours
  Another objective of the trial (only patients undergoing elective radical prostatectomy) is to measure the effect of hydroxyethyl starch on u-Kim1 and u-LFABP, which are also biomarkers of nephrotoxicity
FENa, u-ENaCβ, CH2O, u-AQP2,u-NCC, u-NK2CC | 2-4 hours
  Secondarily to measure the effect of hydroxyethyl starch on the renal tubular transport of sodium and water during elective radical prostatectomy
PRC, p-Ang-II, p -Aldo, p-ANP,P-GDP, p-AVP, p-Endot | 2-4 hours
  Thirdly to measure the effect of hydroxyethyl starch on vasoactive hormones during elective radical prostatectomy
SBP, DBP, heartrate | 2-4 hours
  Fourthly to measure the effect of hydroxyethyl starch on central hemodynamics during elective radical prostatectomy

CONTACTS AND LOCATIONS:
Overall Officials: Anne Sophie P. Kancir, MD PhD, Principal Investigator — Holstebro Regional Hospital
Locations (1):
- Medicinsk forskningsafsnit, Regionshospitalet Holstebro, Holstebro, Denmark

REFERENCES:
- [Derived] Kancir ASP, Johansen JK, Ekeloef NP, Pedersen EB. The effect of 6% hydroxyethyl starch 130/0.4 on renal function, arterial blood pressure, and vasoactive hormones during radical prostatectomy: a randomized controlled trial. Anesth Analg. 2015 Mar;120(3):608-618. doi: 10.1213/ANE.0000000000000596. PMID 25627076